CLINICAL TRIAL: NCT06068062
Title: Implementing OSCE in Team Based Learning Format for Teaching Clinical Skills to Undergraduate Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HITEC-Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ayesha Akram, Associate professor, HITEC-Institute of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: HITECIMS
Record Dates: First submitted 2023-09-26; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: OSCE (Objective Structured Clinical Examination); TBL (Team Based Learning); Teaching Clinical Skills to Undergraduate Medical Students

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Control group (Group A) undergo traditional teaching of skills as routinely carried out in gynecology department during clinical clerkship of three weeks.
- Experimental group (Experimental): Group B undergo intervention in the form of learning session where OSCE will be implemented on principles of Team-based learning.
  Interventions: Other: modification of OSCE using TBL format

INTERVENTIONS:
Other: modification of OSCE using TBL format — Modification of Team-based learning format and implementing OSCE using that modified format to teach clinical skills to medical students.To teach clinical skills this structure of TBL was modified and with use of OSCE following strategy was planned as intervention. First of all, the students were provided with the resource material regarding the skills to be taught. Then a formative OSCE session was organized where students were divided into groups each with 5 students. They were rotated in two OSCE stations. First each student one by one was supposed to perform the task that was clearly documented and was evaluated by peers and facilitator. Immediate feedback from peers and facilitators was given to each student. Students were also instructed to discuss among themselves and designate roles also to make a plan and act like team in performing task on OSCE station 2.
  Arms: Experimental group

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of using OSCE(objective structured clinical exam) on principles of TBL (team based learning) in teaching clinical skills to undergraduate medical students. The main question it aims to answer is whether using OSCE on TBL format is an effective role for teaching clinical skills in undergraduate medical students.

4th year MBBS students included in study after informed written consent. By simple random sampling students divided into two groups i.e. Experimental and control group.

Control group was named Group A while the interventional group was Group B. Control group (Group A) underwent traditional teaching of skills as routinely carried out in gynecology department during clinical clerkship of three weeks. Group B underwent intervention in the form of learning session where OSCE was implemented on principles of Team-based learning. Both groups had pre-test at start of study in the form of two OSCE stations with pre-validated checklists, to check their baseline knowledge. Post-test on same stations was taken after traditional teaching for group A and intervention for group B. The groups were later crossed over so no student was devoid of the learning experience.

ELIGIBILITY:
Inclusion Criteria:

* Willing students of 4th year MBBS HITEC-IMS Taxila who passed their professional exam

Exclusion Criteria:

* • Dropouts and students not willing to participate

  * Students who failed in professional exam and have to appear in supplementary exam.

Ages: 23 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Scores of OSCE stations | 4 weeks (at the end of intervention for experimental group and at the end of clerkship for control group
  post test scores at two OSCE stations (higher post test scores would mean better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Akram, MBBS,FCPS, Principal Investigator — Assistant Professor Gynae/Obs
Locations (1):
- Hitec-Ims, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
OSCE checklists, content validity